CLINICAL TRIAL: NCT00933400
Title: Randomized Controlled Study of a Rapid "Rule Out" Strategy Using Computed Tomography Coronary Angiogram (CTCA) Versus Traditional Care for Low- to Intermediate-Risk Emergency Department (ED) Patients With Potential Acute Coronary Syndromes (ACS)
Brief Title: Computed Tomography Coronary Angiogram (CTCA) Versus Traditional Care in Emergency Department Assessment of Potential Acute Coronary Syndromes (ACS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American College of Radiology (Other)
Collaborators: Pennsylvania Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ACRIN PA 4005
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Results first posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Chest Pain; Acute Coronary Syndrome; Acute Myocardial Infarction; Coronary Artery Disease
Keywords: Computed Tomography; CT Angiography (CTA); Cardiac CT; CT; Cardiac CTA (CCTA); Chest Pain; Heart Attack; Emergency Department; Myocardial Infarction; Cost Effectiveness; Acute Coronary Event; Heart Imaging
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome; Coronary Artery Disease; Myocardial Infarction; Emergencies | interventions — Computed Tomography Angiography; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional Strategy [Group A] (Active Comparator): In the traditional-care arm (Group A:Standard of Care (SOC)), all management and disposition decisions will be made by the healthcare providers caring for the participant. Participants will receive disposition (admit to hospital, admit to cardiac diagnostic unit, or discharge to home), diagnostic testing (none, stress testing, or cardiac catheterization), and treatment according to the team caring for the participant.
  Interventions: Procedure: Traditional Strategy
- CT Coronary Angiography (CTCA)[Group B] (Experimental): In the study CT coronary angiography-based rapid "rule out" arm (Group B), participants will receive initial cardiac troponin and creatinine tests. Upon return of normal laboratory values (including a calculated creatinine clearance), the participants will receive a CT coronary angiography an estimated 90 minutes or as soon as the CT scanner is available following the initial values assessment. Participants with negative test results will be discharged unless other indications for admission per standard of care and follow up will comprise telephone interviews 30 days and 1 year after triage/presentation. Participants with positive test results will be admitted to the hospital for further management as dictated by the admitting team.
  Interventions: Diagnostic Test: CT Coronary Angiography (CTCA)

INTERVENTIONS:
Diagnostic Test: CT Coronary Angiography (CTCA) — CT coronary angiography will be performed without and with contrast in participants randomized to receive imaging as well as traditional care. (For applicable purposes, the decision to perform contrast-enhanced imaging in the presence of a large amount of calcium should be made according to procedures at each individual site.) The imaging test will be considered positive if the participant has a greater than 50% stenosis of the right coronary, left main, left anterior descending, or circumflex arteries or of their branches in contrast-enhanced CT coronary angiography. Results will be communicated to the responsible ED and treating staff immediately upon interpretation; ED staff will determine appropriate course of management. Negative results will result in patient discharge.
  Other Names: CT angiography (CTA); CTCA
  Arms: CT Coronary Angiography (CTCA)[Group B]
Procedure: Traditional Strategy — Participants randomized to traditional care will be assessed and discharged/treated according to routine standard-of-care procedures in the institution's emergency department.
  Other Names: Standard of Care (SOC); Traditional, Standard of Care; Routine Care
  Arms: Traditional Strategy [Group A]

SUMMARY:
This multi-center, randomized, controlled trial conducted in Emergency Departments (ED) compares computed tomography (CT) coronary angiography with the traditional approach (usual care) for low- to intermediate-risk chest pain patients. The primary objective is to estimate the rate of major cardiac events (heart attack or cardiac death) within 30 days in trial participants in Group B who were not found to have significant coronary artery disease by CT coronary angiography. Additional evaluations will comprise health care utilization assessments, including length of hospital stay and re-admissions, cost analysis, and 1-year post-triage/presentation major cardiac event rates.

DETAILED DESCRIPTION:
In this study, participants with potential ACS will be randomized to traditional "rule out" care (Group A) or to traditional care plus CT coronary angiography (Group B) in a ratio of 1:2 traditional versus traditional plus CT coronary angiography.

In Group A, all management and disposition decisions will be made by the healthcare providers caring for the participant. Participants will be admitted to hospital, admitted to cardiac diagnostic unit, or discharged to home. Diagnostic testing and treatment will be decided by the team caring for the participant. Follow up will comprise telephone interviews after 30 days and 1 year from triage/presentation.

In Group B, participants will receive initial cardiac troponin and creatinine blood tests. Upon return of normal laboratory values, the participants will receive a CT coronary angiography an estimated 90 minutes after the initial values assessment or as soon as the CT scanner is available. Participants with negative test results will be discharged; follow up will comprise telephone interviews after 30 days and 1 year from triage/presentation. Participants with positive test results will be admitted to the hospital for further management dictated by the admitting team.

ELIGIBILITY:
Inclusion Criteria:

* Participant is 30 years of age or older
* Participant presents with complaints consistent with potential ACS (e.g., chest pain, shortness of breath, other)
* Participant requires admission or objective testing to exclude ACS
* Participant with initial ECG result without acute ischemia
* Participant with an initial Thrombolysis in Myocardial Infarction (TIMI) Risk Score of 0 to 2
* Participant is willing to provide a written informed consent

Exclusion Criteria:

* Patients who present with symptoms that are clearly not cardiac in origin (e.g., chest pain secondary to herpes zoster, obvious pneumonia, or recent trauma);
* Patients with no initial ECG performed in the ED
* Patients with ST-elevation myocardial infarction (STEMI)
* Patients with existing co-morbidity that requires admission regardless of presence of ACS (e.g., uncontrolled diabetes)
* Patients with known contraindications to CT coronary angiography: Iodinated contrast allergic-like reaction
* Patients who are known to have had CT coronary angiography in the year prior to presentation
* Patients who are known to have normal catheterization results (no or minimal, < 25%, stenosis) in the year prior to presentation
* Patients who are pregnant
* Patients with known renal insufficiency (e.g., creatinine clearance < 60 mL/min/1.73 m2)
* Patients with no telephone or cell phone numbers (preventing follow up)
* Patients unwilling to provide a written informed consent

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1392 (Actual)
Dates: Start 2009-07; Primary Completion 2012-02 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harold I Litt, PhD, Study Chair — University of Pennsylvania Health System
Locations (5):
- United States (5):
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Penn State Hershey - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Penn-Presbyterian Medical Center, Philadelphia, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Bittner DO, Mayrhofer T, Bamberg F, Hallett TR, Janjua S, Addison D, Nagurney JT, Udelson JE, Lu MT, Truong QA, Woodard PK, Hollander JE, Miller C, Chang AM, Singh H, Litt H, Hoffmann U, Ferencik M. Impact of Coronary Calcification on Clinical Management in Patients With Acute Chest Pain. Circ Cardiovasc Imaging. 2017 May;10(5):e005893. doi: 10.1161/CIRCIMAGING.116.005893. PMID 28487318
- [Derived] Litt HI, Gatsonis C, Snyder B, Singh H, Miller CD, Entrikin DW, Leaming JM, Gavin LJ, Pacella CB, Hollander JE. CT angiography for safe discharge of patients with possible acute coronary syndromes. N Engl J Med. 2012 Apr 12;366(15):1393-403. doi: 10.1056/NEJMoa1201163. Epub 2012 Mar 26. PMID 22449295

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited patients presenting to the emergency department (ED) with potential acute coronary syndromes. After the initial electrocardiogram, consenting subjects were randomization to CCTA or traditional care (2:1ratio). Subjects subsequently found to have a creatinine clearance less than 60 ml/minute or who received a pulmonary embolism protocol CT rather than a CCTA were removed from the study.
Groups:
- CT Coronary Angiography (Group B:CCTA): In the study Coronary computed tomographic angiography (CCTA) -based rapid "rule out" arm (Group B), participants will receive initial cardiac troponin and creatinine tests. Upon return of normal laboratory values (including a calculated creatinine clearance), the participants will receive a CT coronary angiography an estimated 90 minutes or as soon as the CT scanner is available following the initial values assessment. Participants with negative test results will be discharged unless other indications for admission per standard of care and follow up will comprise telephone interviews 30 days and 1 year after triage/presentation. Participants with positive test results will be admitted to the hospital for further management as dictated by the admitting team.
- Traditional Strategy (Group A): In the traditional-care arm (Group A), all management and disposition decisions will be made by the healthcare providers caring for the participant. Participants will receive disposition (admit to hospital, admit to cardiac diagnostic unit, or discharge to home), diagnostic testing (none, stress testing, or cardiac catheterization), and treatment according to the team caring for the participant.
Period: Overall Study
Arm/Group | CT Coronary Angiography (Group B:CCTA) | Traditional Strategy (Group A)
Started | 929 | 463
Index Visit | 908 | 462
CCTA Performed | 767 | 0
Vital Status Available 30 Days Post ED Triage | 908 | 462
30 Day Post ED Triage Follow-up Data | 898 | 457
1-year Post ED Triage Follow-up Data | 907 | 461
Completed | 908 | 462
Not Completed | 21 | 1
Not completed — Withdrawal by Subject | 21 | 1

BASELINE CHARACTERISTICS:
Groups:
- CT Coronary Angiography-based Rapid "Rule Out" Arm (Group B): Participants receive initial cardiac troponin/creatinine tests. Upon return of normal laboratory values (including a calculated creatinine clearance), participants receive a CT coronary angiography an estimated 90 minutes or as soon as the CT scanner is available following the initial values assessment. Participants with negative test results will be discharged unless other indications for admission per standard of care and follow up will comprise telephone interviews 30 days and 1 year after triage/presentation. Participants with positive test results will be admitted to the hospital for further management as dictated by the admitting team.
  CT Coronary Angiography(CTCA): CT coronary angiography will be performed without and with contrast in participants randomized to receive imaging as well as traditional care. (For applicable purposes, the decision to perform contrast-enhanced imaging in the presence of a large amount of calcium should be made according to procedures at each individual site.) The imaging test will be considered positive if the participant has a greater than 50% stenosis of the right coronary, left main, left anterior descending, or circumflex arteries or of their branches in contrast-enhanced CT coronary angiography. Results will be communicated to the responsible Emergency Department (ED) and treating staff immediately upon interpretation; ED staff will determine appropriate course of management. Negative results will result in patient discharge.
- Traditional Strategy (Group A): In the traditional-care arm (Group A), all management and disposition decisions will be made by the healthcare providers caring for the participant. Participants will receive disposition (admit to hospital, admit to cardiac diagnostic unit, or discharge to home), diagnostic testing (none, stress testing, or cardiac catheterization), and treatment according to the team caring for the participant.
  Traditional Strategy: Participants randomized to traditional care will be assessed and discharged/treated according to routine standard-of-care (SOC) procedures in the institution's emergency department (ED).
- Total: Total of all reporting groups
Arm/Group | CT Coronary Angiography-based Rapid "Rule Out" Arm (Group B) | Traditional Strategy (Group A) | Total
Number analyzed (Participants) | 908 | 462 | 1370
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (8.9) | 50 (9.5) | 49 (9.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 443 | 202 | 645
  Male | 465 | 260 | 725
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 11 | 32
  Not Hispanic or Latino | 867 | 439 | 1306
  Unknown or Not Reported | 20 | 12 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 11 | 7 | 18
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 520 | 286 | 806
  White | 359 | 158 | 517
  More than one race | 5 | 4 | 9
  Unknown or Not Reported | 9 | 4 | 13
Cardiac history and risk factors [Count of Participants; unit: Participants] — Values represent the number of participants presenting with the specified condition
  Participants
    Hypertension | 463 | 232 | 695
    Hypercholesterolemia | 249 | 118 | 367
    Family History of CAD | 268 | 126 | 394
    Diabetes Mellitus | 130 | 64 | 194
    Current Tobacco use | 291 | 156 | 447
    Cocaine use in last week | 49 | 20 | 69
    Myocardial infarction | 10 | 6 | 16
    Heart failure | 10 | 9 | 19
Presenting electrocardiogram [Count of Participants; unit: Participants] — Randomization occurred after an initial electrocardiogram and results (Normal v non-normal) are presented here
  Participants
    Normal | 584 | 299 | 883
    Nonspecific | 208 | 111 | 319
    Early repolarization | 24 | 14 | 38
    Non-diagnostic | 68 | 24 | 92
    Ischemia (inadequate blood supply) known to be old | 11 | 6 | 17
    Ischemia (inadequate blood supply) not known to be old | 10 | 7 | 17
    ST Elevation consistent with Acute Myocardial Infarction (AMI)-old | 2 | 0 | 2
    Other/Unknown | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Rates of Major Cardiac Events (AMI or Cardiac Death) Within 30 Days
Description: To estimate the rate of major cardiac events (AMI or cardiac death) within 30 days of discharge from Emergency Department (ED) - patient follow-up included telephone interviews 30 days and 1 year after triage/presentation.
  Participants in Group B who were found not to have stenosis of the main or first order coronary branches greater than or equal to 50% by CT coronary angiography were considered negative and considered discharged if they were not designated to receive an inpatient bed or formal observation status.
  All myocardial infarctions were reviewed by an Adjudication Committee to confirm diagnosis.
Time Frame: up to 30 days of discharge from the ED
Measure: Count of Participants; unit: Participants
Groups:
- CT Coronary Angiography (Group B): Participants randomized to CT coronary angiography with scan planned as soon as the CT scanner is available following the initial values assessment (expected within 90 minutes). Participants with negative test results will be discharged unless other indications for admission per standard of care. Participants with positive test results will be admitted to the hospital for further management as dictated by the admitting team.
  CT Coronary Angiography: CT coronary angiography was performed without and with contrast in participants randomized to receive imaging as well as traditional care. (For applicable purposes, the decision to perform contrast-enhanced imaging in the presence of a large amount of calcium should be made according to procedures at each individual site.) The imaging test was considered positive if the participant has a greater than 50% stenosis of the right coronary, left main, left anterior descending, or circumflex arteries or of their branches in contrast-enhanced CT coronary angiography. Results were communicated to the responsible Emergency Department (ED) and treating staff immediately upon interpretation; ED staff will determine appropriate course of management.
- Traditional Strategy (Group A): In the traditional-care arm (Group A), all management and disposition decisions will be made by the healthcare providers caring for the participant. Participants will receive disposition (admit to hospital, admit to cardiac diagnostic unit, or discharge to home), diagnostic testing (none, stress testing, or cardiac catheterization), and treatment according to the team caring for the participant.
  Traditional Strategy: Participants randomized to traditional care will be assessed and discharged/treated according to routine standard-of-care procedures in the institution's emergency department.
- Negative CT Coronary Angiography-based Rapid "Rule Out" (Group B): This group contains only those subjects from Group B where the imaging test was completed and negative: the participant had a <= 50% stenosis of the right coronary, left main, left anterior descending, and circumflex arteries and of their branches in contrast-enhanced CT coronary angiography.
Arm/Group | CT Coronary Angiography (Group B) | Traditional Strategy (Group A) | Negative CT Coronary Angiography-based Rapid "Rule Out" (Group B)
Number analyzed (Participants) | 908 | 462 | 640
Participants
  Death | 0 | 0 | 0
  AMI | 10 | 5 | 0
Statistical Analysis 1: Comparison: CT Coronary Angiography (Group B) vs Traditional Strategy (Group A); Difference in AMI rate. NULL: equal rates of AMI in both Groups; Test type: Equivalence — equivalence margin = 0; Percent Difference = 0.02, 95% CI 2-sided [-5.6 to 5.7]

2. Secondary Outcome: Significant Coronary Artery Disease Detected Within Index Hospitalization as Assessed by Medical Record Review.
Description: The algorithm used for diagnosis of Significant coronary artery disease is provided in the Appendix of the protocol.
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Groups:
- CT Coronary Angiography-based Rapid "Rule Out" (Group B): Participants will receive initial cardiac troponin and creatinine tests. Upon return of normal laboratory values (including a calculated creatinine clearance), the participants will receive a CT coronary angiography an estimated 90 minutes or as soon as the CT scanner is available following the initial values assessment. Participants with negative test results will be discharged unless other indications for admission per standard of care and follow up will comprise telephone interviews 30 days and 1 year after triage/presentation. Participants with positive test results will be admitted to the hospital for further management as dictated by the admitting team.
  CT Coronary Angiography: CT coronary angiography will be performed without and with contrast in participants randomized to receive imaging as well as traditional care. (For applicable purposes, the decision to perform contrast-enhanced imaging in the presence of a large amount of calcium should be made according to procedures at each individual site.) The imaging test will be considered positive if the participant has a greater than 50% stenosis of the right coronary, left main, left anterior descending, or circumflex arteries or of their branches in contrast-enhanced CT coronary angiography. Results will be communicated to the responsible ED and treating staff immediately upon interpretation; ED staff will determine appropriate course of management. Negative results will result in patient discharge.
Arm/Group | CT Coronary Angiography-based Rapid "Rule Out" (Group B) | Traditional Strategy (Group A)
Number analyzed (Participants) | 908 | 462
Participants
  Discharge from ED | 450 | 105
  Admission/observation to ED | 458 | 357
  Significant coronary disease | 82 | 16
Statistical Analysis 1: Comparison: CT Coronary Angiography-based Rapid "Rule Out" (Group B) vs Traditional Strategy (Group A); Difference in Discharge rates. H0: equal rates of Discharge in both Groups; Test type: Equivalence — equivalence margin = 0; Difference (rates) = 26.8, 95% CI 2-sided [21.4 to 32.2]
Statistical Analysis 2: Comparison: CT Coronary Angiography-based Rapid "Rule Out" (Group B) vs Traditional Strategy (Group A); Difference in diagnosis rate of Significant coronary disease at index visit. H0: equal rates in both Groups; Test type: Equivalence — equivalence margin = 0; Difference (percents) = 5.6, 95% CI 2-sided [0.0 to 11.2] — exact procedures were used to estimate and compare rates of detection for significant coronary disease

3. Secondary Outcome: Mean Length of Hospital Stay After Initial Visit
Description: Compare the length of hospital stay in hours between the groups
Time Frame: 1-7 days
Population: Results report for all patient and for those with a negative index visit assessment.
Measure: Mean (Inter-Quartile Range); unit: hours
Arm/Group | CT Coronary Angiography-based Rapid "Rule Out" (Group B) | Traditional Strategy (Group A)
Number analyzed (Participants) | 908 | 462
hours
  Overall | 18.0 [7.6 to 27.2] | 24.8 [19.2 to 30.5]
  Subjects with negative test: number analyzed (Participants) | 681 | 264
  Subjects with negative test | 12.3 [7.0 to 24.3] | 24.7 [19.7 to 29.6]

4. Secondary Outcome: Health Care Utilization During the Index Hospitalization.
Description: Downstream diagnostic test during the index visit including Hospital admission or observation.
Time Frame: 1-7 Days
Measure: Count of Participants; unit: Participants
Arm/Group | CT Coronary Angiography-based Rapid "Rule Out" (Group B) | Traditional Strategy (Group A)
Number analyzed (Participants) | 908 | 462
Participants
  CCTA | 767 | 26
  Stress testing, with or without imaging | 124 | 267
  Cardiac catheterization | 37 | 18
  No additional Diagnostic tests | 80 | 167
  Hosp. Admission or observation | 458 | 357
Statistical Analysis 1: Comparison: CT Coronary Angiography-based Rapid "Rule Out" (Group B) vs Traditional Strategy (Group A); H0: no difference in Patient disposition (Discharge) rates between arms; Test type: Superiority; binomial proportion = 26.8, 95% CI 2-sided [21.4 to 32.2] — Exact confidence intervals for the difference in proportions

5. Secondary Outcome: Cardiac Health Care Utilization 1 Year Post Triage/Presentation.
Time Frame: Through 1-yr study follow up
Population: Subjects with index visit and know outcome at 1-yr post ED triage
Measure: Count of Participants; unit: Participants
Groups:
- CT Coronary Angiography-based Rapid "Rule Out" Arm (Group B): Participants will receive initial cardiac troponin and creatinine tests. Upon return of normal laboratory values (including a calculated creatinine clearance), the participants will receive a CT coronary angiography an estimated 90 minutes or as soon as the CT scanner is available following the initial values assessment. Participants with negative test results will be discharged unless other indications for admission per standard of care and follow up will comprise telephone interviews 30 days and 1 year after triage/presentation. Participants with positive test results will be admitted to the hospital for further management as dictated by the admitting team.
  CT Coronary Angiography: CT coronary angiography will be performed without and with contrast in participants randomized to receive imaging as well as traditional care. (For applicable purposes, the decision to perform contrast-enhanced imaging in the presence of a large amount of calcium should be made according to procedures at each individual site.) The imaging test will be considered positive if the participant has a greater than 50% stenosis of the right coronary, left main, left anterior descending, or circumflex arteries or of their branches in contrast-enhanced CT coronary angiography. Results will be communicated to the responsible ED and treating staff immediately upon interpretation; ED staff will determine appropriate course of management. Negative results will result in patient discharge.
Arm/Group | CT Coronary Angiography-based Rapid "Rule Out" Arm (Group B) | Traditional Strategy (Group A)
Number analyzed (Participants) | 852 | 438
Participants
  Emergency department visit | 305 | 166
  Hospital admission: number analyzed (Participants) | 843 | 432
  Hospital admission | 137 | 74
  Cardiologist office visit: number analyzed (Participants) | 821 | 423
  Cardiologist office visit | 148 | 53
  CCTA: number analyzed (Participants) | 822 | 422
  CCTA | 2 | 5
  Stress testing without imaging: number analyzed (Participants) | 827 | 424
  Stress testing without imaging | 19 | 2
  Stress testing with imaging: number analyzed (Participants) | 824 | 422
  Stress testing with imaging | 60 | 33
  Catheterization: number analyzed (Participants) | 829 | 423
  Catheterization | 24 | 13
  Echocardiogram: number analyzed (Participants) | 824 | 425
  Echocardiogram | 49 | 26

6. Secondary Outcome: Major Adverse Cardiac Event (MACE, Including Myocardial Infarction & Cardiac Death) and Revascularization for Participants Within 1 Year Post Triage/Presentation
Description: MACE at 1 year was determined by Patient telephone contact Medical record review Records at the presenting and neighboring hospitals were reviewed for repeat visits When these methods failed to provide survival information, we searched the Social Security Death Master File
Time Frame: Through 1-yr study follow up
Population: Subject with index visit, Vital status available at 1-yr post ED triage, and known outcome
Measure: Count of Participants; unit: Participants
Arm/Group | CT Coronary Angiography-based Rapid "Rule Out" (Group B) | Traditional Strategy (Group A)
Number analyzed (Participants) | 907 | 461
Participants
  All-Cause Mortality | 2 | 3
  Cardiac Death: number analyzed (Participants) | 906 | 460
  Cardiac Death | 1 | 0
  AMI: number analyzed (Participants) | 870 | 444
  AMI | 11 | 5
  MACE: number analyzed (Participants) | 870 | 443
  MACE | 12 | 5
  Revascularization: number analyzed (Participants) | 872 | 444
  Revascularization | 25 | 7
Statistical Analysis 1: Comparison: CT Coronary Angiography-based Rapid "Rule Out" (Group B) vs Traditional Strategy (Group A); Compare all cause mortality between groups; Test type: Equivalence — The trial was powered to test the principal hypothesis that the major adverse cardiac event (MACE, including myocardial infarction and cardiac death) rate among patients found not to have significant CAD on CCTA exceeds 1%; binomial proportion = -0.4, 95% CI 2-sided [-6.0 to 5.2] — Exact confidence intervals for the difference in proportions
Statistical Analysis 2: Comparison: CT Coronary Angiography-based Rapid "Rule Out" (Group B) vs Traditional Strategy (Group A); Compare Cardiac Death between groups; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; binomial proportion = 0.1, 95% CI 2-sided [-5.5 to 5.7] — Exact confidence intervals for the difference in proportions
Statistical Analysis 3: Comparison: CT Coronary Angiography-based Rapid "Rule Out" (Group B) vs Traditional Strategy (Group A); Compare AMI between groups; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; binomial proportion = 0.1, 95% CI 2-sided [-5.6 to 5.9] — Exact confidence intervals for the difference in proportions
Statistical Analysis 4: Comparison: CT Coronary Angiography-based Rapid "Rule Out" (Group B) vs Traditional Strategy (Group A); Compare MACE between groups; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; binomial proportion = 03, 95% CI 2-sided [-5.5 to 6.0] — Exact confidence intervals for the difference in proportions
Statistical Analysis 5: Comparison: CT Coronary Angiography-based Rapid "Rule Out" (Group B) vs Traditional Strategy (Group A); Compare Revascularization between groups; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; binomial proportion = 1.3, 95% CI 2-sided [-4.4 to 7.0] — Exact confidence intervals for the difference in proportions

ADVERSE EVENTS:
Time Frame: within 30 days of study scan and at 1 year follow up (or study termination visit if occurring prior to 1 year follow up)
Description: Adverse events were assessed via record review, patient and secondary contacts, and the Social Security Death Master File was consulted for vital status (date last accessed for all patients, January 25, 2012).
Arm/Group | CT Coronary Angiography-based Rapid "Rule Out" (Group B) | Traditional Strategy (Group A)
All-Cause Mortality (participants affected / at risk) | 2/929 | 3/463
Serious Adverse Events (participants affected / at risk) | 0/929 | 2/463
Other Adverse Events (participants affected / at risk) | 0/929 | 0/463
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CT Coronary Angiography-based Rapid "Rule Out" (Group B) (N=929) | Traditional Strategy (Group A) (N=463)
General disorders and administration site conditions (death) (General disorders) | 0 (0) | 1 (1) — 10011914 - self-inflicted gunshot wound to the head (per Death certificate)
10040741 - Sinus Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) — Pt had a CCTA as part of the usual care arm. Unclear whether bradycardia was result of IV dye or beta- blocker

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2010-03-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT00933400/Prot_SAP_ICF_000.pdf